CLINICAL TRIAL: NCT00263211
Title: The Impact Of Platelet Function Inhibition On Circulating Cancer Cells In Metastatic Breast Cancer Patients
Brief Title: A Study of the Effects of Inhibiting Platelet Function on Circulating Cancer Cells in Breast Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped due to low percentage of patients with detectable CTCs at baseline.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-0427 / 201107340
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Metastatic; Platelet
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plavix and Aspirin (Experimental): Patients will receive a 300 mg loading dose of Plavix on day 1, followed by 75 mg/day, and aspirin 81 mg per day starting day 1. Treatment will be continued until the treating physician elects to resume systemic therapy for the treatment of breast cancer or until unacceptable toxicity is observed. A pill diary will be collected monthly to monitor patients' compliance with the medication regimen.
  Interventions: Drug: Plavix; Drug: Aspirin
- Observation only (No Intervention): Observation by treating physician

INTERVENTIONS:
Drug: Plavix
  Other Names: Clopidogrel Bisulfate
  Arms: Plavix and Aspirin
Drug: Aspirin
  Other Names: acetylsalicylic acid
  Arms: Plavix and Aspirin

SUMMARY:
The purpose of this study is to determine the effects of Plavix and aspirin in women with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women with metastatic breast cancer who are completing planned course of chemotherapy with planned treatment break
* On stable hormone therapy for at least 2 months are also eligible for the study
* Estimated survival of at least 3 months
* No platelet inhibitor therapy within 1 month of study entry
* Platelets ≥ 100,000
* Coagulation screening tests within normal range (INR between 0.81 and 1.20)
* Normal kidney and liver function as defined by:

  * Aspartate aminotransferase(AST)/serum glutamic oxaloacetic transaminase (SGOT))/alanine aminotransferase(ALT) ≤ 2 x Institutional Normal
  * Creatinine ≤ 2 x Institutional Normal
* Able to provide signed, informed consent.

Exclusion Criteria:

* Patients going on to surgery
* Patients with a serious bleeding disorder that make them inappropriate candidates for NSAID therapy
* Patients with history of significant bleeding related to peptic ulcer disease
* Patients on standing doses of NSAIDS or platelet function inhibitors
* Patients on standing doses of anti-coagulants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine N Weilbaecher, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened for enrollment in January 6, 2006 and closed enrollment in May 25, 2010
Period: Overall Study
Arm/Group | Plavix and Aspirin | Observation Only
Started | 24 | 24
Completed | 19 | 23
Not Completed | 5 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Disease Progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plavix and Aspirin | Observation Only | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (12.01) | 58.4 (12.06) | 55.79 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48
The Number of Participants with Detectable Positive Circulating Tumor Cells (CTCs=>1) at Baseline [Number; unit: participants] — The number of participants with detectable CTCs (>= 1 CTC) was calculated at baseline.
  participants | 12 | 18 | 30
Human Epidermal Growth Factor Receptor 2 Positivity (HER2+) [Number; unit: participants] — Some breast cancers have high amounts of a protein called HER2/neu on the surface of the cancer cells (called HER2/neu-positive (HER2-positive) breast cancer). The HER2/neu protein is important for cancer cell growth.
  participants | 8 | 10 | 18
Estrogen Receptor Positivity (ER+) [Number; unit: participants] — Estrogen Receptor + means that the breast cancer is considered "hormone-receptor-positive."
  participants | 15 | 13 | 28
Number of Metastatic Sites [Number; unit: participants]
  1 | 8 | 9 | 17
  2 | 7 | 7 | 14
  ≥3 | 9 | 8 | 17
Number of Previous Metastatic Chemotherapy Regimens [Number; unit: participants]
  0 | 6 | 4 | 10
  1 | 5 | 8 | 13
  2 | 4 | 6 | 10
  ≥3 | 9 | 6 | 15
Number of Previous Metastatic Endocrine Therapies [Number; unit: participants]
  0 | 8 | 11 | 19
  1 | 7 | 3 | 10
  ≥2 | 9 | 10 | 19
Number of Participants Concurrently using Trastuzumab [Number; unit: participants] | 5 | 9 | 14
Number of Participants Concurrently using Bisphosphonate [Number; unit: participants] | 12 | 9 | 21
Number of Participants who Smoke [Number; unit: participants] | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Platelet Inhibition of Circulating Tumor Cells (CTCs) Measured by the Number of Patients With Detectable CTCs
Description: Measured by number of patients who have detectable circulating tumor cells
Time Frame: Week 4
Population: Plavix & Aspirin arm has 19 evaluable patients. 5 withdrew before 1-month data collection: death n=1 and withdrawal of consent n=1 prior to starting; surgery plans n=1; patient preference n=1; platelet inhibition use n=1; Observation only arm had 23 evaluable patients ; 1 patient withdrew during the first month due to disease progression.
Measure: Number; unit: participants
Arm/Group | Plavix and Aspirin | Observation Only
Number analyzed (Participants) | 19 | 23
participants | 11 | 15

2. Primary Outcome: Safety and Tolerability of Aspirin and Plavix Measured by the Number of Patients Who Discontinue the Study Drug
Description: Measured by number of patients who discontinue administration of study drug because of toxicity and the incidence categorized by type.
Time Frame: Maximum of 6 months
Population: Plavix and Aspirin: 1 patient withdrew consent prior to starting 1 patient died prior to starting
Measure: Number; unit: participants
Arm/Group | Plavix and Aspirin | Observation Only
Number analyzed (Participants) | 22 | 24
participants
  Bleeding (possibly related) | 1 | 0
  Back pain (unlikely related) | 1 | 0

3. Secondary Outcome: Percentage of Patients With a Given Absolute Number of Circulating Tumor Cells (Broken Into Categories) Plotted Against Time
Description: Percent of patients with a given number/range of CTCs ( 0, 1-5 >+ 5) vs. time baseline 2-weeks and 1 month for plavix & Aspirin arm and observation only
Time Frame: Baseline, 2 weeks and 1 month
Population: Denominator for Plavix & Aspirin arm at Baseline=22, at 2 weeks =20, at 4 weeks =19 Denominator for Observation only at Baseline=24, at 2 weeks=19, at 4 weeks =23
Measure: Number; unit: percentage of participants
Arm/Group | Plavix and Aspirin | Observation Only
Number analyzed (Participants) | 22 | 24
percentage of participants
  Baseline 0 CTCs | 40.00 | 22.73
  2 week 0 CTCs | 45.00 | 40.00
  1 month 0 CTCs | 41.18 | 35.00
  Baseline 1-5 CTCs | 45.00 | 63.64
  2 weeks 1-5 CTCs | 31.58 | 45.00
  1 month 1-5 CTCs | 52.94 | 55.00
  Baseline >=5 CTS | 15.00 | 13.64
  2 weeks >=5 CTCs | 21.05 | 15.00
  1 month >=5 CTCs | 5.88 | 10.00

4. Secondary Outcome: Mean Aspirin-Mediated Platelet Inhibition vs. Time Plotted for Plavix and Aspirin and Observation Groups
Description: Mean platelet inhibition vs. time plotted for Plavix & Aspirin Arm and Observation group. Citrated whole blood is added to a test carriage containing fibrinogen-coated beads and a platelet activator (arachidonic acid to synthesize thromboxane A2). Using a turbidimetric-based optical detection system, aggregation of activated platelets to fibrinogen-coated beads increase light transmittance which is reported in Aspirin Reaction Units (ARU).
Time Frame: Baseline, 2 weeks and 1 month
Population: Denominator for Plavix & Aspirin arm baseline n=22, 2 weeks n=20, 1 month n=19 Denominator for Observation only arm baseline n=24 , 2-weeks n=19, 1 month n=23
Measure: Mean (Standard Deviation); unit: Aspirin Reaction Units
Arm/Group | Plavix and Aspirin | Observation Only
Number analyzed (Participants) | 22 | 24
Aspirin Reaction Units
  Baseline Aspirin Reaction UnitsARU | 610.39 (57.64) | 579.81 (92.10)
  2 weeks ARU | 435.33 (56.50) | 578.35 (151.10)
  1 month ARU | 455.44 (94.70) | 593.58 (88.81)

5. Secondary Outcome: Clopidogrel-Mediated Percent of Platelet Inhibition vs. Time Plotted for Aspirin and Plavix and Observation Groups
Description: Mean Clopidogrel-Mediated platelet inhibition (% inhibition) vs. time for Aspirin and Plavix and Observation groups
Time Frame: Baseline, 2 weeks and 1 month
Population: Mean Platelet inhibition Denominator for Plavix & Aspirin arm baseline n=22, 2 weeks n=20, 1 month n=19 Denominator for control group baseline n=24 , 2-weeks n=19, 1 month n=23
Measure: Mean (Standard Deviation); unit: percentage of platelet inhibition
Arm/Group | Plavix and Aspirin | Observation Only
Number analyzed (Participants) | 22 | 24
percentage of platelet inhibition
  Baseline | 9.85 (16.13) | 13.00 (21.93)
  2 weeks | 37.35 (30.38) | 9.05 (7.96)
  1 month | 35.56 (30.90) | 7.05 (7.07)

6. Secondary Outcome: Progression Free Survival
Time Frame: Maximum of 6 months
Population: This trial was terminated early due to futility, subjects were not followed for progression free-survival.
Groups:
- Plavix and Aspirin: Patients will receive a 300 mg loading dose of Plavix on day 1, followed by 75 mg/day, and aspirin 81 mg per day starting day 1. Treatment will be continued until the treating physician elects to resume systemic therapy for the treatment of breast cancer or until unacceptable toxicity is observed. A pill diary will be collected monthly to monitor patients' compliance with the medication regimen.
  Plavix
Arm/Group | Plavix and Aspirin | Observation Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Plavix and Aspirin | Observation Only
Serious Adverse Events (participants affected / at risk) | 3/24 | 1/24
Other Adverse Events (participants affected / at risk) | 24/24 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plavix and Aspirin (N=24) | Observation Only (N=24)
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Edema (Blood and lymphatic system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Calf Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Mucositis (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plavix and Aspirin (N=24) | Observation Only (N=24)
ALT (Investigations) | 4 | 0
AST (Investigations) | 1 | 0
Albumin, serum low (Metabolism and nutrition disorders) | 0 | 1
Alkaline Phosphate (Investigations) | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 2
Bruising (Injury, poisoning and procedural complications) | 9 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Lymphedema (Vascular disorders) | 0 | 2
Dermatology other-Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatology other-bilateral breast inflammation and discoloration and alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 2
Dizziness (Nervous system disorders) | 6 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Edema: Limb (General disorders) | 5 | 5
Edema Head and Neck (General disorders) | 0 | 1
Edema Trunk/genital (General disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 8 | 8
Fever (General disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 3
Hematoma (Vascular disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 7 | 7
Hemorrhage Respiratory Nose (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hemorrhage, GU Vagina (Reproductive system and breast disorders) | 1 | 0
Hot Flashes (Vascular disorders) | 4 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Infection G 1/2 Normal ANC Pulmonary (Neck NOS) (Infections and infestations) | 1 | 0
Infection G 1/2 Normal Pulmonary (upper airway) (Infections and infestations) | 0 | 1
Infection Unknown ANC Auditory /ear (external) (Infections and infestations) | 1 | 0
Infection Unknown ANC Pulmonary (Pharynx) (Infections and infestations) | 0 | 1
Infection Unknown ANC Renal (Urinary tract) (Infections and infestations) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 3
Joint -function (Musculoskeletal and connective tissue disorders) | 1 | 0
Leukocytes (Investigations) | 6 | 6
Lymphatic other swelling (General disorders) | 0 | 1
Lymphopenia (Investigations) | 5 | 5
Metabolic Lab/ Other BUN high (Metabolism and nutrition disorders) | 0 | 3
Plasma protein low (Metabolism and nutrition disorders) | 3 | 0
Mood Alteration-Anxiety (Psychiatric disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 8 | 9
Neuropathy -cranial motor face (Nervous system disorders) | 0 | 1
Neuropathy -motor (Nervous system disorders) | 1 | 0
Neuropathy Sensory (Nervous system disorders) | 6 | 6
Neutrophils (Investigations) | 3 | 3
PTT (Investigations) | 0 | 2
Pain Neuralgia/Neuropathy (Nervous system disorders) | 0 | 2
Pain GI (Abdomen NOS) (Gastrointestinal disorders) | 2 | 2
Pain GI (stomach) (Gastrointestinal disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint Pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Muscle Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 8 | 8
Hip and Jaw Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain Pulmonary (Chest Thorax NOS) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Platelets (Investigations) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash acne/acneiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Rash dermatitis assoc. with reaction : chemo (Skin and subcutaneous tissue disorders) | 1 | 0
Rash desquamation (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Renal (Slight blood in urine/hematuria) (Renal and urinary disorders) | 2 | 0
Rigors/chills (General disorders) | 0 | 1
Persistent vaginal herpes (Reproductive system and breast disorders) | 1 | 0
Skin Breakdown decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Sweating (General disorders) | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Urine color change (Renal and urinary disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 4
Heartburn (Gastrointestinal disorders) | 0 | 3
Liver Pain (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Inclusion of patients with no or few CTC's limited ability to distinguish anti-platelet therapeutic effect.

Early termination because of low probability of reaching statistical significance for primary outcome

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No